CLINICAL TRIAL: NCT02912754
Title: A Phase I/II Trial of Ruxolitinib in Chronic Lymphocytic Leukemia Patients at Risk for Progression on Ibrutinib
Brief Title: Ruxolitinib Combined With Ibrutinib in Chronic Lymphocytic Leukemia Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dr. David Spaner, Clinical Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424XCA05T
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2016-09

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ruxolitinib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibrutinib plus Ruxolitinib (Experimental): Patients taking ibrutinib for relapsed CLL will add ruxolitinib twice per day at the dose identified in a preliminary phase I trial for 7 cycles (3 weeks on/2 weeks off).
  Interventions: Drug: ruxolitinib; Drug: ibrutinib
- Ibrutinib alone (No Intervention): Patients will continue to take Ibrutinib for the equivalent period of time.

INTERVENTIONS:
Drug: ruxolitinib — ruxolitinib will be added to ibrutinib or 3 out of 5 weeks per cycle
  Other Names: jakafi
  Arms: Ibrutinib plus Ruxolitinib
Drug: ibrutinib — patients will be taking ibrutinib for at least 6 months and will continue to take it at the same dose and schedule while taking ruxolitinib
  Other Names: imbruvica
  Arms: Ibrutinib plus Ruxolitinib

SUMMARY:
This study involves adding the kinase inhibitor Ruxolitinib to Ibrutinib to treat Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
Ibrutinib is an effective drug that can extend the lives of CLL patients but it is not curative as a single agent and may eventually select for more aggressive disease. Survival of CLL cells in the presence of Ibrutinib may be enabled by signals from the microenvironment where the leukemia cells originate. These signals are transmitted into the cells by Janus Kinases (JAKs) such as janus kinase 1 (JAK1) and janus kinase 2 (JAK2). According, JAK inhibitors may overcome the cytoprotective properties of the CLL microenvironment and help to improve outcomes with Ibrutinib.

The JAK2 inhibitor Ruxolitinib is licensed for use in myelofibrosis and polycythemia rubra vera and its toxicity and efficacy as a single agent in CLL has been studied in two previous clinical trials. As a single agent, Ruxolitinib was inferior to Ibrutinib. However, Ruxolitinib was shown to cooperate with Ibrutinib and increase killing of CLL cells in vitro. Based on these observations, it is hypothesized that Ruxolitinib will significantly improve the therapeutic efficacy of single-agent Ibrutinib.

This is a single center phase I/II trial to determine the efficacy and safety of ruxolitinib tablets in CLL patients being treated until progression with Ibrutinib and considered at risk to progress on the basis of persistent lymphocytosis and lymphadenopathy after 1 year of Ibrutinib or elevated beta-2-microglobulin (b2M) levels after 6 months of Ibrutinib. Ruxolitinib will be administered for 21 days of a 35-day cycle to be repeated 6 more times.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL meeting published diagnostic criteria.
2. CLL currently being treated with Ibrutinib due to relapsed/refractory disease or primary del17p cytogenetic lesions at a daily dose of 420 mg and:

   * failure of plasma b2M levels to decrease below 2.5 mg/L after 6 months after starting Ibrutinib.
   * persistent lymphocytosis (>5x106 cells/L) and splenomegaly or lymphadenopathy (marker node >1.5 cm on CT scans) after 1 year of taking Ibrutinib.
3. Not currently treated with other agents for CLL.
4. Serum bilirubin, and alanine transferase less than or equal to twice the upper limit of normal.
5. Platelets >75x109/L. Absolute neutrophil count (ANC)>.75x109/L. Hemoglobin greater than or equal to 65 g/L
6. Age >18 years old
7. Eastern Cooperative Oncology Group (ECOG) < 2

Exclusion Criteria:

1. Patients with inadequate bone marrow reserve at baseline visit as demonstrated by at least one of the following: a. ANC<.75x109/L b. platelets <75x109/L without the assistance of growth factors, thrombopoietic factors, or platelet transfusions. C. hemoglobin <65 g/L despite transfusions.
2. Patients who have or have had progressive multifocal leukoencephalopathy (PML).
3. Patients with clinically significant bacterial, fungal, parasitic or viral infection, which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
4. Patients with known active hepatitis A, B, C or who are HIV-positive or who are at risk for hepatitis B virus (HBV) reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care prior to alloSCT that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
5. Primary immunodeficiency such as X-linked agammaglobulinemia or common variable immunodeficiency.
6. Patients with active and inactive ('latent') tuberculosis infection.
7. Involvement of the central nervous system by lymphoma or leukemia.
8. Richter's transformation or prolymphocytic leukemia.
9. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
10. Use of glucocorticoids above the equivalent of 10 mg of prednisone daily within 4 weeks prior to treatment.
11. Major surgery within 4 weeks prior to treatment.
12. Patients with a history of malignancy in the past 3 years except for treated, early-stage squamous or basal cell carcinoma.
13. History or current diagnosis of uncontrolled or significant cardiac disease, including any of the following: a. myocardial infarction within last 6 months. b. uncontrolled congestive heart failure. c. unstable angina within last 6 months. d. exertional angina. e. clinically significant (symptomatic) cardiac arrhythmias (eg. bradyarrhythmias, sustained ventricular tachycardia, and clinically significant second or third degree block without a pacemaker).
14. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
15. Renal failure requiring dialysis or serum creatinine >176.8 microM and patients with moderate (creatinine clearance of 30-50 ml/min) and severe (creatinine clearance<30 ml/min) renal impairment with platelet counts less than 100,000/ml.
16. Patients with mild, moderate, or severe hepatic impairment or inadequate liver function defined by any of direct bilirubin, alanine amino transferase (ALT), or aspartate aminotransferase (AST)>2.5 x upper limit of normal (ULN).
17. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral ruxolitinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
18. Patients with known hypersensitivity to ruxolitinib or other JAK1/2 inhibitors, or to their excipients.
19. Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 30 days of screening or 5 half-lives (whichever is longer) prior to the first dose of study drug.
20. Significant concurrent, uncontrolled medical condition which, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
21. Subjects who are unable to comprehend or are unwilling to sign an informed consent form (ICF).
22. Sexually active males who do not agree to use condoms during intercourse while taking ruxolitinib and for 3 months after stopping treatment (N.B. the mean elimination half-life of ruxolitinib is around 3 hours) and not father a child in this period. Vasectomized men must also agree to use a condom during intercourse to prevent delivery of ruxolitinib via seminal fluid.
23. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human choriogonadotropin (HCG) laboratory test (>5 mIU/ml).
24. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study duration inclusive of 30 day safety follow up. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. Incase of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). the vasectomized male partner should be the sole partner for that subject.
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
25. Use of strong CYP3A4 inhibitors for patients in the phase I component of the trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of ruxolitinib in combination with Ibrutinib. | 2 years
  identify the MTD of ruxolitinib with ibrutinib

SECONDARY OUTCOMES:
ability of Ruxolitinib to increase the depth of response to Ibrutinib | 2 years
  identify the number of complete responses that occur when ruxolitinib is added to ibrutinib

OTHER OUTCOMES:
effect of Ruxolitinib on levels of plasma cytokines and chemokines | 3 years
  quantification of plasma cytokines and chemokines

CONTACTS AND LOCATIONS:
Overall Officials: David E Spaner, MD, Principal Investigator — Sunnybrook Odette Cancer Center
Locations (1):
- Sunnybrook Odette Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
the results from the study will be published in peer-review journals

REFERENCES:
- [Result] Oppermann S, Lam AJ, Tung S, Shi Y, McCaw L, Wang G, Ylanko J, Leber B, Andrews D, Spaner DE. Janus and PI3-kinases mediate glucocorticoid resistance in activated chronic leukemia cells. Oncotarget. 2016 Nov 8;7(45):72608-72621. doi: 10.18632/oncotarget.11618. PMID 27579615
- [Result] Spaner DE, Wang G, McCaw L, Li Y, Disperati P, Cussen MA, Shi Y. Activity of the Janus kinase inhibitor ruxolitinib in chronic lymphocytic leukemia: results of a phase II trial. Haematologica. 2016 May;101(5):e192-5. doi: 10.3324/haematol.2015.135418. Epub 2016 Jan 27. No abstract available. PMID 26819050
- [Derived] Xia M, Luo TY, Shi Y, Wang G, Tsui H, Harari D, Spaner DE. Effect of Ibrutinib on the IFN Response of Chronic Lymphocytic Leukemia Cells. J Immunol. 2020 Nov 15;205(10):2629-2639. doi: 10.4049/jimmunol.2000478. Epub 2020 Oct 16. PMID 33067379
- [Derived] Spaner DE, McCaw L, Wang G, Tsui H, Shi Y. Persistent janus kinase-signaling in chronic lymphocytic leukemia patients on ibrutinib: Results of a phase I trial. Cancer Med. 2019 Apr;8(4):1540-1550. doi: 10.1002/cam4.2042. Epub 2019 Mar 7. PMID 30843659
- [Derived] Shi Y, Wang G, Muhowski EM, McCaw L, Wang C, Bjarnason G, Woyach JA, Spaner DE. Ibrutinib reprograms the glucocorticoid receptor in chronic lymphocytic leukemia cells. Leukemia. 2019 Jul;33(7):1650-1662. doi: 10.1038/s41375-019-0381-4. Epub 2019 Jan 29. PMID 30696950